CLINICAL TRIAL: NCT05538039
Title: Comparison of the Effectiveness of Two Different Distraction Interventions in Reducing Preoperative Anxiety of Children and Parents Who Are Scheduled for Elective Surgery: A Randomized Controlled Study
Brief Title: Reducing Anxiety of Children and Their Parents in the Pre-elective Surgery Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta University of Applied Sciences (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IspartaUAS
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Preoperative Care; Child; Parent; Anxiety
Keywords: Preoperative Care; Child; Parents; Nursing care; Randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Distract with play dough (Experimental): The intervention will begin approximately 30 minutes before premedication. The initiative will be applied to both the child and the parent participating in the research. Attempts to distract with play dough will be conducted under investigative coaching for at least 10 minutes. If after 10 minutes the child or parent wants to continue playing, they will be told that they can play as long as they want. Each family will be given 4 boxes of play dough. After the play is played, the play dough will not be put back in the package, and the child and parents will be told that they can keep the shapes they have made if they wish. The play dough used will be provided by the researchers and will be given to the participants after the intervention.
  Interventions: Other: Distract with play dough
- Distract with play kaleidoscope (Experimental): The intervention will begin approximately 30 minutes before premedication. The initiative will be applied to both the child and the parent participating in the research. Attempts to distract with the kaleidoscope will be conducted under investigative coaching for at least 10 minutes. It is a game tool that reproduces the outside image when viewed from inside the kaleidoscope. This image is obtained thanks to the glasses placed inside the kaleidoscope at different angles, and the images change as the kaleidoscope is rotated. If after 10 minutes the child or parent wants to continue playing, they will be told that they can play as long as they want. Each child and parent will be given a separate kaleidoscope.
  Interventions: Other: Distract with play kaleidoscope
- Control Group (Other): The participants in the control group will be given routine nursing care.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Distract with play dough — Distract with play dough
  Arms: Distract with play dough
Other: Distract with play kaleidoscope — Distract with play kaleidoscope
  Arms: Distract with play kaleidoscope
Other: Control group — Routine nursing care
  Arms: Control Group

SUMMARY:
It is emphasized in the studies that the child and parent anxiety that occurs in pediatric surgery should be prevented or reduced. According to previous studies, one way to reduce child and parent anxiety in the preoperative process is distraction interventions the child and family with preoperative family-centered activities. Teaching children anxiety coping skills with the involvement of their parents can reduce preoperative anxiety. This study was planned to Comparison of the effectiveness of two different distraction interventions (distraction with play dough- distraction with kaleidoscope) in reducing preoperative anxiety of children and parents who are scheduled for elective surgery

DETAILED DESCRIPTION:
Aim: This study was planned to Comparison of the effectiveness of two different distraction interventions (distraction with play dough- distraction with kaleidoscope) in reducing preoperative anxiety of children and parents who are scheduled for elective surgery

Method: This study was planned as a randomized controlled trial. The sample of the study will consist of 105 children aged 5-12, who will be operated on at Akdeniz University Hospital, and their parents. Randomization result; It was planned to include a total of 105 children and their parents in 3 groups: distraction with play dough group (intervention group 1)= 35, distraction with kaleidoscope group (intervention group 2)= 35 , and control group= 35 children and parents.

Child and parent information form will be used to collect data, Modified Yale Preoperative Anxiety Scale will be used to collect data in child sample, and Spielberger State Anxiety Scale will be used to collect data in parent sample.

Intervention and Data Collection: Randomization will be performed after the purpose of the study is explained to the child and parent who agreed to participate in the study and after obtaining consent. Immediately after the pre-test (first measurement) is given to the children assigned to intervention group 1 and their parents, attempts to distract attention with play dough will be applied for 10 minutes. If they wish, the child and parents will be told that they can continue to play with the play dough until premedication. Children assigned to intervention group 2 and their parents will be distracted with a kaleidoscope for 10 minutes immediately after the pre-test (first measurement) is done. If they wish, the child and parents will be told that they can continue to play with the kaleidoscope until premedication. Participants randomized to the control group will be given routine standard nursing care. The second measurement will be administered 15 minutes after the interventions (before premedication=post test), and the control group 25 minutes after the first measurement (before premedication=posttest). Thus, the effectiveness of the initiatives and their comparison with each other will be evaluated.

The data of the research will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The process of evaluating the data will be carried out with the support of a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Being a child between the ages of 5 and 12 who is planned for elective surgery
* Being the parent of a 5-12 year old child scheduled for elective surgery
* Child and parent have no vision, hearing or speech problems
* Child and parent do not have a mental or neurological disability
* The child and parents do not have an anxiety disorder
* Child and parent can speak and understand Turkish

Exclusion Criteria:

* Change in surgical operation date
* Using another distraction technique

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Reducing children's pre-operative anxiety | Anxiety levels of children will be evaluated twice. The first measurement will be made 30 minutes before the premedication, and the last measurement will be made just before the premedication.
  The decrease in anxiety levels of children whose attention is diverted with play dough and kaleidoscope is an outcome measure. This reduction will be measured with the "Modified Yale Preoperative Anxiety Scale". Outcome criteria will be evaluated twice, approximately 30 minutes before premedication and immediately before premedication (pretest-posttest) in the Pediatric Surgery Service. The scale consists of twenty-two items and five categories. Each category gets one point out of four. The higher the score on the scale, the greater the anxiety. In the post-test, it will be evaluated whether there is a decrease according to the pre-test score. Statistical significance will be set to p < 0.05.
Reducing parent's pre-operative anxiety | Anxiety levels of parents will be evaluated twice. The first measurement will be made 30 minutes before the premedication, and the last measurement will be made just before the premedication.
  The decrease in anxiety levels of parents of children whose attention is diverted with play dough and kaleidoscope is an outcome measure. This decrease will be measured by the "Spielberger State Anxiety Scale". Outcome criteria will be evaluated twice in Pediatric Surgery Service, approximately 30 minutes before premedication and just before premedication (pretest-posttest). The 4-point Likert-type scale, consisting of 20 items in total, measures the anxiety of the person at a certain time. For scores above 42 points, it indicates a high level of anxiety. In the post-test, it will be evaluated whether there is a decrease according to the pre-test score. Statistical significance will be set to p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Fahriye RN PAZARCIKCI, PhD, Study Director — Isparta University of Applied Sciences; Fatma RN TIRAŞ, Study Chair — Akdeniz University; Şevkiye RN DİKMEN, Study Chair — Akdeniz University; Emine RN EFE, Professor, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Aytekin A, Doru O, Kucukoglu S. The Effects of Distraction on Preoperative Anxiety Level in Children. J Perianesth Nurs. 2016 Feb;31(1):56-62. doi: 10.1016/j.jopan.2014.11.016. Epub 2015 Nov 11. PMID 26847781
- [Background] Bulut M, Kucuk Alemdar D, Bulut A, Salci G. The Effect of Music Therapy, Hand Massage, and Kaleidoscope Usage on Postoperative Nausea and Vomiting, Pain, Fear, and Stress in Children: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Dec;35(6):649-657. doi: 10.1016/j.jopan.2020.03.013. Epub 2020 Jul 20. PMID 32703758
- [Background] Dwairej DA, Obeidat HM, Aloweidi AS. Video game distraction and anesthesia mask practice reduces children's preoperative anxiety: A randomized clinical trial. J Spec Pediatr Nurs. 2020 Jan;25(1):e12272. doi: 10.1111/jspn.12272. Epub 2019 Oct 1. PMID 31576651
- [Background] Stewart B, Cazzell MA, Pearcy T. Single-Blinded Randomized Controlled Study on Use of Interactive Distraction Versus Oral Midazolam to Reduce Pediatric Preoperative Anxiety, Emergence Delirium, and Postanesthesia Length of Stay. J Perianesth Nurs. 2019 Jun;34(3):567-575. doi: 10.1016/j.jopan.2018.08.004. Epub 2018 Nov 7. PMID 30413359